CLINICAL TRIAL: NCT07267299
Title: Efficacy of Switching Participants Treated With Restasis to TRYPTYR
Brief Title: Switching From Restasis to TRYPTYR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006763-Restasis
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Eye Diseases; Chronic Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases

STUDY DESIGN:
Intervention Model Description: Switching to acoltremon 0.003% will significantly improve the signs and symptoms of participants who were being treated with Restasis at 28 days post-treatment compared to baseline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- acoltremon 0.003%. (Experimental): Switching to acoltremon 0.003% will significantly improve the signs and symptoms of participants who were being treated with Restasis at 28 days post-treatment compared to baseline.
  Interventions: Drug: acoltremon 0.003%

INTERVENTIONS:
Drug: acoltremon 0.003% — Participants who are using restasis will be switched to acoltremon 0.003%

SUMMARY:
Switching to acoltremon 0.003% will significantly improve the signs and symptoms of participants who were being treated with Restasis at 28 days post-treatment compared to baseline. Dry eye disease (DED) is a prevalent condition that commonly affects patients of working age in addition to the elderly. DED is a complex condition that results in ocular symptoms such as dryness and burning and signs such as decreased tear production (aqueous deficient DED) or increased tear evaporation (evaporative DED). Unfortunately, there is not a perfect correlation between DED signs and symptoms, which makes diagnosis and timely treatment challenging.

DETAILED DESCRIPTION:
Acoltremon 0.003% was recently approved by the US Food and Drug Administration (FDA) as the first transient receptor potential melastatin 8 (TRPM8) agonist for the treatment of DED.9, 10 Acoltremon acts by activating TRPM8 receptors expressed on the neurons of the ophthalmic division of the trigeminal nerve, which is the nerve that innervates the cornea and eyelid.9 This drugs subsequently modulates cold thermoreceptor to increase tear production and promote a cooling sensation, which promotes symptomatic relief. While acoltremon 0.003% has been significantly shown to improve the signs and symptoms of DED patient, the community currently lacks data describing how patients who are being treated with Restasis (cyclosporine ophthalmic emulsion), yet are not having their expectations met with the drug, respond to being switched to acoltremon 0.003%. These data are important because they could demonstrate that a DED drug with a different mechanism of action can still be effective when another treatment does not meet the patient's expectations. Thus, the purpose of this study is to determine if acoltremon 0.003% can significantly improve the signs and symptoms of DED suffers who are not currently being successfully treated with Restasis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Have a history of DED for at least the past 6 months.
* Are currently using Restasis as directed by their eye care provider for ≥1 month.
* Participant intends to stop Restasis in the near future because and expressed dissatisfaction with effectiveness of Restasis in reducing dry eye symptoms..
* Are symptomatic as determined with the Eye Dryness visual analog scale (VAS) (Score ≥50), SPEED (≥7), and have an abnormal Schirmer test score [≥2 to <10 mm/5 min]) at Screening/Baseline.
* Have corrected distance visual acuity of 20/100 or better.
* Willing to discontinue contact lens wear throughout the study.

Exclusion Criteria:

* Have a systemic health condition that is known to alter tear film physiology (e.g., primary and secondary Sjögren's syndrome).
* Have a history of ocular surgery within the past 12 months.
* Have a history of severe ocular trauma, active ocular infection or inflammation that is not dry eye related.
* Punctal plugs in place for < 3 months and/or Lacrifill in place for > 5 months.
* Have ever used Accutane or are currently using ocular medications (must washout from all dry eye medications/treatments at least 1 week before entry, except for Restasis).
* Use of artificial tears within 2 hours prior to the baseline visit or during the study.
* Are pregnant or breast feeding.
* Have had a physical meibomian gland treatment withing 1 month of enrollment.
* Have a condition or be in a situation, which in the investigator's opinion, may put the participant at significant risk, may confound the results, or may significantly interfere with their study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Change between pre- and post-drop in unanesthetized Schirmer test score on Day 1 | 1 day
  schirmers strip wetting/time will be measured between pre and post drop. With quicker wetting with greater voulme being considered better.

SECONDARY OUTCOMES:
Change in SPEED scores | 28 days
  participants will complete the standardized speed questionnaire at baseline and at 28 days. To determine improvement, lower speed scores are considered better.
Change in SPEED scores | 14 days
  participants will complete the standardized speed questionnaire at baseline and at 14 days. To determine improvement, lower speed scores are considered better.